CLINICAL TRIAL: NCT06411795
Title: Rectus Sheath Block With Liposomal Bupivacaine Versus Thoracic Epidural Analgesia for Pain Control Following Pancreatoduodenectomy: A Prospective, Randomized, Non-Inferiority Trial
Brief Title: Rectus Sheath Block With Liposomal Bupivacaine Versus Thoracic Epidural Analgesia for Pain Control Following Pancreatoduodenectomy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ANES-2023-31918; NCI-2024-02287 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ANES-2023-31918 (Other: University of Minnesota/Masonic Cancer Center); P30CA077598 (NIH)
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Duodenal Neoplasm; Pancreatic Neoplasm
MeSH Terms: conditions — Duodenal Neoplasms; Pancreatic Neoplasms | interventions — Bupivacaine; Hydromorphone; Iopamidol; Tea; High-Energy Shock Waves; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Patients and providers will not be blinded to the analgesic technique
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group E (TEA) (Experimental): Prior to pancreatoduodenectomy, patients undergo thoracic epidural placement and receive bupivacaine and hydromorphone continuous infusion via epidural for up to 72 hours postoperatively. Patients also receive iopamidol via epidural and undergo x-ray imaging on study.
  Interventions: Drug: Bupivacaine; Drug: Hydromorphone; Drug: Iopamidol; Other: Medical Chart Review; Other: Questionnaire Administration; Drug: Thoracic Epidural Analgesia; Procedure: X-Ray Imaging
- Group RS (rectus sheath block) (Experimental): Prior to pancreatoduodenectomy, patients undergo ultrasound and receive bupivacaine and liposomal bupivacaine injection into the rectus sheath.
  Interventions: Drug: Bupivacaine; Drug: Liposomal Bupivacaine; Other: Medical Chart Review; Other: Questionnaire Administration; Procedure: Ultrasound Imaging

INTERVENTIONS:
Drug: Bupivacaine — Given via epidural and injection
  Other Names: AH 250
Drug: Hydromorphone — Given via epidural
  Other Names: (-)-Hydromorphone; Dihydromorphinone; Hydromorphon
  Arms: Group E (TEA)
Drug: Iopamidol — Given via epidural
  Other Names: Isovue; Niopam; Solutrast
  Arms: Group E (TEA)
Drug: Liposomal Bupivacaine — Given injection
  Other Names: Bupivacaine Liposome Injectable Suspension; Exparel
  Arms: Group RS (rectus sheath block)
Other: Medical Chart Review — Ancillary studies
  Other Names: Chart Review
Other: Questionnaire Administration — Ancillary studies
Drug: Thoracic Epidural Analgesia — Undergo thoracic epidural placement
  Other Names: TEA; Thoracic Epidural
  Arms: Group E (TEA)
Procedure: Ultrasound Imaging — Undergo ultrasound
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US
  Arms: Group RS (rectus sheath block)
Procedure: X-Ray Imaging — Undergo x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray
  Arms: Group E (TEA)

SUMMARY:
This phase II trial compares the effect of rectus sheath block with liposomal bupivacaine to thoracic epidural analgesia (TEA) on pain control in patients following surgical removal of all or part of the pancreas and duodenectomy (pancreatoduodenectomy). Administering long acting local anesthetics, such as liposomal bupivacaine, in between the muscle layers of the abdomen (rectus sheath block) may help with pain relief during and after surgery. TEA uses a needle to insert a flexible plastic catheter into the thoracic spine to administer anesthetic and pain medication, such as bupivacaine and hydromorphone, to treat pain in the thoracic and upper abdominal areas during and after surgery. Epidurals have been successfully used to treat pain after surgery, however, it does have a risk of low blood pressure which may limit the use in the thoracic approach. Rectus sheath blocks with liposomal bupivacaine may be as effective as TEA in reducing pain in patients following a pancreatoduodenectomy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if rectus sheath blocks with liposomal bupivacaine provide non-inferior analgesia compared with thoracic epidural analgesia (TEA) for patients undergoing pancreatoduodenectomy.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP EPIDURAL (E): Prior to pancreatoduodenectomy, patients undergo thoracic epidural placement and receive bupivacaine and hydromorphone continuous infusion via epidural for up to 72 hours postoperatively. Patients also receive iopamidol via epidural and undergo x-ray imaging on study.

GROUP RECTUS SHEATH (RS): Prior to pancreatoduodenectomy, patients undergo ultrasound and receive bupivacaine and liposomal bupivacaine injection into the rectus sheath.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age 18 and older, undergoing open pancreaticoduodenectomy at the University of Minnesota will be included in the study

Exclusion Criteria:

* Patients with contraindication to block placement (coagulopathy, local anesthetic allergy, infection)
* Patients with chronic opioid use (at least 30 milligram morphine equivalents [MME] for 3 or more weeks leading up to surgery)
* Patients unable to understand the quality of recovery survey intellectual barriers. This will be determined by the primary investigator/attending anesthesiologist's discretion
* Patient refusal and those who have opted out of research
* Pregnant patients - will be assessed through review of the medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Milligram morphine equivalents (MME) | Up to 96 hours after open pancreatoduodenectomy
  Opioid consumption will be evaluated as a non-inferiority hypothesis using a two-sample t-test to compare the groups, with the conclusion of statistical significance being drawn from the corresponding confidence interval for the differences in mean MMEs between groups.

SECONDARY OUTCOMES:
Pain scores | At 24, 48, 72 and 96 hours
  Pain scores at rest and with movement will be assessed using a numeric rating scale pain scores where 0 is no pain and 10 is worst pain.
Hospital length of stay | Up to 7 days after surgery
  Average hospital length of stay
Opioid consumption | 96 hours
  Average Opioid consumption (milligrams)
Time to return of bowel function | Up to 7 days after surgery
  Average time to return of bowel function will be measured by first oral intake.
Incidence of nausea, vomiting, hypotension and pruritis | At 24 hours, 48 hours, 72 hours and 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: James Flaherty, Principal Investigator — University of Minnesota Masonic Cancer Center
Locations (1):
- University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota, United States